CLINICAL TRIAL: NCT01070342
Title: Methodological Improvement in Measuring Efficacy Outcome in Antihypertensive Trials in Children
Brief Title: Ambulatory Blood Pressure Monitoring in Children
Acronym: ABPM
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: University of California, San Diego (Other); Arkansas Children's Hospital Research Institute (Other); University of Cincinnati (Other); University of Louisville (Other)
Responsible Party: Sponsor
Other Study IDs: CTSAP1; ULI-RR024989 (Other Grant/Funding Number: National Center for Research Resources)
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chidren ages 6 to 18: Children ages 6 to 18 years will be available for participation in this multicenter study. Subjects will be enrolled from community based general pediatric clinics and other well-child care areas within participating hospitals and clinics of the four participating sites. Enrollment will continue until a total of 85 subjects from each age category (6-<12 years and ≥12- <18 years) successfully complete the study.
  Interventions: Device: Spacelabs 90217

INTERVENTIONS:
Device: Spacelabs 90217 — Comparison of the two ways to measure blood pressure: using the ambulatory blood pressure device (Spacelabs 90217) versus the standard method of measuring blood pressure is done by using a stethoscope and a blood pressure cuff.

SUMMARY:
Ambulatory Blood Pressure Monitoring (ABPM) potentially offers a superior way to screen children for entry into antihypertensive trials, assuring that only those with true hypertension are enrolled.10 In addition, ABPM offers a better method to measure response to drug therapy.11-16 The ABPM device most commonly used in children (Spacelabs 90217 - Issaquah, Washington) has not been independently validated for use in this population. In 1993, the British Hypertension Society (BHS) published a protocol for validating ABPM devices, including guidance for validation studies in children.17 More recently, the Working Group on Blood Pressure Monitoring of the European Society of Hypertension published revisions to these guidelines, but did not include children in this update.18 Unfortunately, the original BHS protocol suggests using a smaller group of children than the protocol outlines for adults. Since BP in children is more variable than in adults, this guidance is unlikely to be adequate for children. Hence, a large, stringent validation study needs to be conducted in a cohort of children using the methods similar to those used to validate the device in adults. Performance of the proposed validation study is needed to allow for the incorporation of ABPM into clinical trial designs of anti-hypertensives in children which will ultimately allow for more accurate identification of the hypertensive population and determination of response to therapy along with allowing for assessment of the chronobiologic profile of drug response over the dosing interval.9

DETAILED DESCRIPTION:
The diagnosis and treatment of hypertension remains a challenge in children and adolescents.1 At present the diagnosis is made during medical encounters and depends on randomly applied auscultatory or oscillometric techniques.2 These measurements are influenced by multiple factors including diurnal variation, stress related effects (most notably the fact that the measurement is being performed in a physician's office or clinic), observer bias and the measurement process itself. In addition, these standard approaches provide little information regarding blood pressure and its variability in the patients' ambient environments.3,4 If and when a diagnosis of hypertension is made, lifestyle changes are often prescribed. In children and adolescents these recommendations meet with mixed results that often frustrate patients and families as well as caregivers. In most cases, where sufficient concern exists regarding the long-term health of end organs such as the heart, kidney, eye and brain, pharmacotherapy is recommended. Unfortunately, in these instances drugs are prescribed with little information to guide proper, age-related dosing or safety assessment. In studies conducted over the last decade more than half of the agents marketed for adults with hypertension failed to demonstrate sufficient activity in children and adolescents to meet regulatory requirements for labeling.5 While a significant amount of this apparent ambiguity appears to be related to the design of the studies assessing the efficacy and safety of these drugs in pediatric patients, perhaps a more significant problem in these studies was the determination of who is actually hypertensive in the first place. This supplement addresses this issue directly by introducing an innovative approach to the diagnosis of hypertension in children and adolescents. Once validated, ambulatory BP monitoring may be used to describe and model the chronobiological patterns of blood pressure among patients who have been recently diagnosed with hypertension using standard clinical criteria. This is a unique opportunity to assess treatment naïve patients and compare an innovative new approach to what is currently the gold standard.

The current project is designed specifically to validate the use of ambulatory blood pressure monitoring (ABPM) in children and adolescents so that it may be used as a clinical tool for unambiguously making the diagnosis of hypertension in this patient population and then be used to guide pharmacotherapeutic intervention. The use of ABPM in children was first documented in 19916 and has subsequently been employed in children as young as 2 months of age. Despite its adjunctive use by more than 60% of pediatric nephrologists in North America, the device currently used in the majority of pediatric practices and research centers has never been validated in a pediatric population.

In contrast, ABPM has become a world-wide standard for monitoring blood pressure in adults with suspected hypertension. It offers the advantages of multiple measurements of a dynamic process over a protracted period of time and permits the evaluation of diurnal patterns and nocturnal disease. It also offers distinct advantages in monitoring patients in their natural environment without observer bias while permitting objective assessment of apparent drug resistance and hypotensive events that might occur on therapy. Finally, ABPM measurements have been demonstrated to better correlate with cardiovascular morbidity and mortality than casual measurements.7 They also correlate with end organ damage in children.8 Performance of the proposed validation study is needed to allow for incorporation of ABPM into clinical trial designs related to the diagnosis and treatment of hypertension in children. ABPM will ultimately allow for more accurate determination of response to therapy and asses the chronobiologic profile of drug response over the dosing interval. Of the devices currently marketed, the Spacelabs 90217 offers the range of cuff sizes required by the pediatric population. Thus, it is this monitor that will be validated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-18 years inclusive.
2. Mid-arm circumference measures 12-50 cm.
3. Informed consent/assent.

Exclusion Criteria:

1. Known AV fistula, unrepaired congenital heart disease, or other anatomical anomaly affecting cardiac output and/or normal cardiac circulation.
2. Cardiac arrhythmias which may prevent the ABPM device from obtaining an accurate blood pressure measurement.
3. Anatomical anomalies preventing measuring blood pressure in the non-dominant arm on multiple occasions.
4. Ingestion of caffeine, tobacco exposure, or strenuous exercise within 30 minutes before study blood pressure measurements.
5. Any condition that in the opinion of the principal investigator would affect the subject's ability to safely and accurately complete all study procedures.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children ages 6 to 18 years will be available for participation in this multicenter study. Subjects will be enrolled from community based general pediatric clinics and other well-child care areas within participating hospitals and clinics of the four participating sites. Enrollment will continue until a total of 85 subjects from each age category (6-<12 years and ≥12- <18 years) successfully complete the study. In addition, enrollment will be dependent upon mean qualifying blood pressure and arm circumference such that a wide range of both are represented in each age group.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To validate the Ambulatory Blood Pressure Monitoring device most commonly used in children (Spacelabs 90217 - Issaquah, Washington) has not been independently validated for use in this population. | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Blumer, Ph.D., M.D., Principal Investigator — Universtiy Hosptials Case Medical Center
Locations (2):
- United States (2):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - University of Louisville Research Foundation, Inc., Louisville, Kentucky

REFERENCES:
- [Background] Whelton PK, Beevers DG, Sonkodi S. Strategies for improvement of awareness, treatment and control of hypertension: results of a panel discussion. J Hum Hypertens. 2004 Aug;18(8):563-5. doi: 10.1038/sj.jhh.1001738. PMID 15116145
- [Background] Park MK, Menard SM. Accuracy of blood pressure measurement by the Dinamap monitor in infants and children. Pediatrics. 1987 Jun;79(6):907-14. PMID 3588145
- [Background] Stergiou GS, Baibas NM, Gantzarou AP, Skeva II, Kalkana CB, Roussias LG, Mountokalakis TD. Reproducibility of home, ambulatory, and clinic blood pressure: implications for the design of trials for the assessment of antihypertensive drug efficacy. Am J Hypertens. 2002 Feb;15(2 Pt 1):101-4. doi: 10.1016/s0895-7061(01)02324-x. PMID 11863243
- [Background] Stergiou GS, Rarra VC, Yiannes NG. Changing relationship between home and office blood pressure with increasing age in children: the Arsakeion School study. Am J Hypertens. 2008 Jan;21(1):41-6. doi: 10.1038/ajh.2007.18. PMID 18271071
- [Background] Benjamin DK Jr, Smith PB, Jadhav P, Gobburu JV, Murphy MD, Hasselblad V, Baker-Smith C, Califf RM, Li JS. Pediatric antihypertensive trial failures: analysis of end points and dose range. Hypertension. 2008 Apr;51(4):834-40. doi: 10.1161/HYPERTENSIONAHA.107.108886. Epub 2008 Mar 10. PMID 18332283
- [Background] Portman RJ, Yetman RJ, West MS. Efficacy of 24-hour ambulatory blood pressure monitoring in children. J Pediatr. 1991 Jun;118(6):842-9. doi: 10.1016/s0022-3476(05)82193-6. PMID 2040918
- [Background] White WB. Importance of aggressive blood pressure lowering when it may matter most. Am J Cardiol. 2007 Aug 6;100(3A):10J-16J. doi: 10.1016/j.amjcard.2007.05.009. Epub 2007 May 25. PMID 17666192
- [Background] Belsha CW, Wells TG, McNiece KL, Seib PM, Plummer JK, Berry PL. Influence of diurnal blood pressure variations on target organ abnormalities in adolescents with mild essential hypertension. Am J Hypertens. 1998 Apr;11(4 Pt 1):410-7. doi: 10.1016/s0895-7061(98)00014-4. PMID 9607378
- [Background] O'Brien E. Dipping comes of age: the importance of nocturnal blood pressure. Hypertension. 2009 Mar;53(3):446-7. doi: 10.1161/HYPERTENSIONAHA.108.127571. Epub 2009 Jan 26. No abstract available. PMID 19171787
- [Background] Urbina E, Alpert B, Flynn J, Hayman L, Harshfield GA, Jacobson M, Mahoney L, McCrindle B, Mietus-Snyder M, Steinberger J, Daniels S; American Heart Association Atherosclerosis, Hypertension, and Obesity in Youth Committee. Ambulatory blood pressure monitoring in children and adolescents: recommendations for standard assessment: a scientific statement from the American Heart Association Atherosclerosis, Hypertension, and Obesity in Youth Committee of the council on cardiovascular disease in the young and the council for high blood pressure research. Hypertension. 2008 Sep;52(3):433-51. doi: 10.1161/HYPERTENSIONAHA.108.190329. Epub 2008 Aug 4. No abstract available. PMID 18678786
- [Background] Weber MA, White WB, Giles TD, Bakris GL, Neutel JM, Smith DH, Davidai G. An effectiveness study comparing algorithm-based antihypertensive therapy with previous treatments using conventional and ambulatory blood pressure measurements. J Clin Hypertens (Greenwich). 2006 Apr;8(4):241-50; quiz 251-2. doi: 10.1111/j.1524-6175.2005.05221.x. PMID 16596026
- [Background] Lacourciere Y, Neutel JM, Schumacher H. Comparison of fixed-dose combinations of telmisartan/hydrochlorothiazide 40/12.5 mg and 80/12.5 mg and a fixed-dose combination of losartan/hydrochlorothiazide 50/12.5 mg in mild to moderate essential hypertension: pooled analysis of two multicenter, prospective, randomized, open-label, blinded-end point (PROBE) trials. Clin Ther. 2005 Nov;27(11):1795-805. doi: 10.1016/j.clinthera.2005.11.014. PMID 16368450
- [Background] Smith DH, Cramer MJ, Neutel JM, Hettiarachchi R, Koval S. Comparison of telmisartan versus losartan: meta-analysis of titration-to-response studies. Blood Press Monit. 2003 Jun;8(3):111-7. doi: 10.1097/00126097-200306000-00004. PMID 12900588
- [Background] Coats AJ. Benefits of ambulatory blood pressure monitoring in the design of antihypertensive drug trials. Blood Press Monit. 1996 Apr;1(2):157-160. PMID 10226219
- [Background] Guthrie R, Reggi DR, Plesher MM, Saini RK, Battikha JP. Efficacy and safety of fosinopril/hydrochlorothiazide combinations on ambulatory blood pressure profiles in hypertension. Fosinopril/Hydrochlorothiazide Investigators. Am J Hypertens. 1996 Apr;9(4 Pt 1):306-11. doi: 10.1016/0895-7061(95)00359-2. PMID 8722432
- [Background] Verdecchia P, Gatteschi C, Benemio G, Boldrini F, Guerrieri M, Porcellati C. Duration of the antihypertensive action of atenolol, enalapril and placebo: a randomized within-patient study using ambulatory blood pressure monitoring. Int J Clin Pharmacol Ther Toxicol. 1988 Nov;26(11):570-4. PMID 2854116
- [Background] O'Brien E, Petrie J, Littler W, de Swiet M, Padfield PL, Altman DG, Bland M, Coats A, Atkins N. An outline of the revised British Hypertension Society protocol for the evaluation of blood pressure measuring devices. J Hypertens. 1993 Jun;11(6):677-9. doi: 10.1097/00004872-199306000-00013. No abstract available. PMID 8397248
- [Background] O'Brien E, Pickering T, Asmar R, Myers M, Parati G, Staessen J, Mengden T, Imai Y, Waeber B, Palatini P, Gerin W; Working Group on Blood Pressure Monitoring of the European Society of Hypertension. Working Group on Blood Pressure Monitoring of the European Society of Hypertension International Protocol for validation of blood pressure measuring devices in adults. Blood Press Monit. 2002 Feb;7(1):3-17. doi: 10.1097/00126097-200202000-00002. No abstract available. PMID 12040236
- [Background] National High Blood Pressure Education Program Working Group on High Blood Pressure in Children and Adolescents. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. Pediatrics. 2004 Aug;114(2 Suppl 4th Report):555-76. No abstract available. PMID 15286277
- [Background] Bland JM, Altman DG. Statistical methods for addressing agreement between measurements. Biochemica Clinica 1987; 11:339-404.
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ; Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Recommendations for blood pressure measurement in humans and experimental animals: Part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Hypertension. 2005 Jan;45(1):142-61. doi: 10.1161/01.HYP.0000150859.47929.8e. Epub 2004 Dec 20. PMID 15611362